CLINICAL TRIAL: NCT02893215
Title: Silent Atrial Fibrillation - Screening of High-risk Groups for Atrial Fibrillation (The Silence Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Valborg Heinesen, MD, Hvidovre University Hospital
Other Study IDs: H-16015331
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heart failure: Screening for silent AF with Zenicor thumb-ECG: Patients older than 65 years, diagnosed with heart failure, without any history of atrial fibrillation, ongoing OAC treatment, implanted device or recent stroke/TIA.
  Interventions: Other: Screening for silent AF with Zenicor thumb-ECG
- Diabetes mellitus II: Screening for silent AF with Zenicor thumb-ECG: Patients older than 65 years, diagnosed with diabetes mellitus II, without any history of atrial fibrillation, ongoing OAC treatment, implanted device or recent stroke/TIA.
  Interventions: Other: Screening for silent AF with Zenicor thumb-ECG

INTERVENTIONS:
Other: Screening for silent AF with Zenicor thumb-ECG — Each patient has a device for 14 days, which monitorizes their heart rhythm. They send the ecg four times daily.
  Other Names: Zenicor Medical Systems

SUMMARY:
The primary aim of the present study is to screen high-risk type 2 diabetes patients and heart failure patients without any history of atrial fibrillation (AF), ongoing oral anticoagulation (OAC) treatment, implanted device or recent stroke/Transient Ischemic Attack (TIA), for silent AF.

Moreover, we aim to establish the prevalence of two or more risk factors for stroke in patients with heart failure and diabetes mellitus type 2 (DM2) with the aim of assessing the feasibility for this group to undergo AF screening.

Overall, the aim of the study is to prevent stroke in high-risk patients groups through identification of silent (asymptomatic) atrial fibrillation.

DETAILED DESCRIPTION:
The number of screened patients with respectively heart failure and type 2 diabetes with a risk score (Congestive Heart Failure, Hypertension, Aged 75 years or older, Diabetes, Stroke / transient cerebral ischemia, Vascular disease, Aged 65 years or older and Sex category (CHADSVASc)) of two or more, the number of these patients excluded due to AF or ongoing AF, the number of eligible patients not included for other reasons, and, finally, number of included patients will be listed.

Patients eligible for screening will be supplied with a hand-held ECG-recorder developed by Zenicor Medical Systems (www.zenicor.com) and will transmit recordings 4 times daily (morning, midday, evening -at meals - and before bedtime) and in case of symptoms, for 14 days.

The transmitted ECGs will be digitally stored, analyzed and screened for AF. All AF episodes will recorded and the day and time of the arrhythmia will be registered.

Eligible patients will be given brief oral and the more thorough written patient information about the study, and offered an appointment for the first meeting, which will happen in the Cardiological out-patient clinic in Copenhagen University Hospital (Hvidovre) with a member of the project group. During the first meeting, the patient will get more information about the study and has the possibility to ask questions. If the patient wants to bring a relative or friend already at this meeting, this can be arranged. If the patient meets the criteria and is interested in participation he/she will be invited to participation in the study. The patient gets the rest of the information material, i.e. written informed consent declaration, and is given a period for questioning and consideration of participation for at least three days. If the patient wants another visit for further information and possibly with participation of a relative or friend, such a visit is scheduled, and the patient can be included at this visit, and written informed consent declaration can be given to the project group member.

Heart failure patients will have a standardized echocardiography and diabetes patients will have supplementary registration of HbA1c, and latest blood glucose value. The latest level of creatinine and creatinine clearance will be registered for all patients (DM2 and congestive heart failure (CHF)).

Every patient is given a Study identification (ID) number and there will be a key file linking this number and the patient ID; thus, the dataset is anonymized.

All ECG's will be analyzed using a soft ware based algorithm which has been developed in order to exclude normal recordings (sinus rhythm without irregularities).

Patients with newly detected AF will be referred to the local cardiology out-patient clinic or if present OAC clinic for treatment according to established guidelines including OAC treatment. Here the patients will be informed about the options of OAC treatment, the reasons why we want to offer it, including the risk of developing cerebral ischemic stroke, precautions with this treatment and the risks connected to OAC treatment. The treatment with OAC is not a part of the screening study.

ELIGIBILITY:
Inclusion Criteria:

* Systolic Congestive Heart Failure diagnosed by echocardiography showing a left ventricular ejection fraction (LVEF) ≤ 40%.
* Diagnosed Diabetes Mellitus type II.
* Age 65 years or older
* CHADS-Vasc (Risk score) 2 or higher

Exclusion Criteria:

* Previous history of AF
* Ongoing OAC treatment
* Implanted device
* Recent stroke/TIA

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with congestive heart failure and without any history of atrial fibrillation, ongoing OAC treatment, implanted device or recent stroke/TIA
  Patients with DM-II and without any history of atrial fibrillation, ongoing OAC treatment, implanted device or recent stroke/TIA
Sampling Method: Non-Probability Sample
Enrollment: 1622 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with silent atrial fibrillation as assessed by handheld ECG measurements in high-risk heart failure patients. | 14 days
Number of participants with silent atrial fibrillation as assessed by handheld ECG measurements in high-risk type 2 diabetes patients. | 14 days

SECONDARY OUTCOMES:
Number of participants with supraventricular ectopic activity. | 14 days
  Supraventricular ectopic activity defined as three supraventricular premature beats or more as assessed by handheld ECG.
Number of participants with micro-atrial fibrillation. | 14 days
  Micro-atrial fibrillation defined as atrial fibrillation shorter than 30 seconds or atrial runs longer than five supraventricular premature beats in a run as assessed by handheld ECG.
Number of participants with high risk of stroke in a heart failure population. | 2 years
  High risk patients defined as patients aged 65 years or older and at least one additional risk score point without known atrial fibrillation or ongoing oral anticoagulation.
Number of participants with high risk of stroke in a type 2 diabetes population. | 2 years
  High risk patients defined as patients aged 65 years or older and at least one additional risk score point without known atrial fibrillation or ongoing oral anticoagulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Dixen, MD, Principal Investigator — Hvidovre University Hospital
Locations (9):
- Austria (3):
  - Department of Cardiology, Krankenhaus der Elisabethinen, Linz
  - Kepler Universitätsklinikum GmbH, Linz
  - Krankenhaus der Barmherzigen Brüder Linz, Linz
- Hvidovre University Hospital, Department of cardiology, Hvidovre, Denmark
- Sweden (5):
  - Bjurholms Hälsocentral, Bjurholm
  - Grytnäs Hälsocentral, Kalix
  - The Karolinske Institute, Department of Cardiology, Danderyd Hospital, Stockholm
  - Ålidhems Hälsocentral, Umeå
  - Vindelns Hälsocentral, Vindeln

IPD SHARING:
Plan to Share IPD: No
The ethical approval do not allow us to share individualised data.

REFERENCES:
- [Background] Kannel WB, Benjamin EJ. Status of the epidemiology of atrial fibrillation. Med Clin North Am. 2008 Jan;92(1):17-40, ix. doi: 10.1016/j.mcna.2007.09.002. PMID 18060995
- [Background] Qvist JF, Sorensen PH, Dixen U. Hospitalisation patterns change over time in patients with atrial fibrillation. Dan Med J. 2014 Jan;61(1):A4765. PMID 24393590
- [Background] Friberg L, Bergfeldt L. Atrial fibrillation prevalence revisited. J Intern Med. 2013 Nov;274(5):461-8. doi: 10.1111/joim.12114. Epub 2013 Aug 7. PMID 23879838
- [Background] Svennberg E, Engdahl J, Al-Khalili F, Friberg L, Frykman V, Rosenqvist M. Mass Screening for Untreated Atrial Fibrillation: The STROKESTOP Study. Circulation. 2015 Jun 23;131(25):2176-84. doi: 10.1161/CIRCULATIONAHA.114.014343. Epub 2015 Apr 24. PMID 25910800
- [Background] Flegel KM, Shipley MJ, Rose G. Risk of stroke in non-rheumatic atrial fibrillation. Lancet. 1987 Mar 7;1(8532):526-9. doi: 10.1016/s0140-6736(87)90174-7. PMID 2881082
- [Background] Wolf PA, Dawber TR, Thomas HE Jr, Kannel WB. Epidemiologic assessment of chronic atrial fibrillation and risk of stroke: the Framingham study. Neurology. 1978 Oct;28(10):973-7. doi: 10.1212/wnl.28.10.973. PMID 570666
- [Background] Friberg L, Hammar N, Rosenqvist M. Stroke in paroxysmal atrial fibrillation: report from the Stockholm Cohort of Atrial Fibrillation. Eur Heart J. 2010 Apr;31(8):967-75. doi: 10.1093/eurheartj/ehn599. Epub 2009 Jan 27. PMID 19176537
- [Background] Hart RG, Pearce LA, Rothbart RM, McAnulty JH, Asinger RW, Halperin JL. Stroke with intermittent atrial fibrillation: incidence and predictors during aspirin therapy. Stroke Prevention in Atrial Fibrillation Investigators. J Am Coll Cardiol. 2000 Jan;35(1):183-7. doi: 10.1016/s0735-1097(99)00489-1. PMID 10636278
- [Background] Savelieva I, Camm AJ. Clinical relevance of silent atrial fibrillation: prevalence, prognosis, quality of life, and management. J Interv Card Electrophysiol. 2000 Jun;4(2):369-82. doi: 10.1023/a:1009823001707. PMID 10936003
- [Background] Rizos T, Wagner A, Jenetzky E, Ringleb PA, Becker R, Hacke W, Veltkamp R. Paroxysmal atrial fibrillation is more prevalent than persistent atrial fibrillation in acute stroke and transient ischemic attack patients. Cerebrovasc Dis. 2011;32(3):276-82. doi: 10.1159/000330348. Epub 2011 Aug 31. PMID 21893980
- [Background] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Background] Glotzer TV, Hellkamp AS, Zimmerman J, Sweeney MO, Yee R, Marinchak R, Cook J, Paraschos A, Love J, Radoslovich G, Lee KL, Lamas GA; MOST Investigators. Atrial high rate episodes detected by pacemaker diagnostics predict death and stroke: report of the Atrial Diagnostics Ancillary Study of the MOde Selection Trial (MOST). Circulation. 2003 Apr 1;107(12):1614-9. doi: 10.1161/01.CIR.0000057981.70380.45. Epub 2003 Mar 24. PMID 12668495
- [Background] Gage BF, Waterman AD, Shannon W, Boechler M, Rich MW, Radford MJ. Validation of clinical classification schemes for predicting stroke: results from the National Registry of Atrial Fibrillation. JAMA. 2001 Jun 13;285(22):2864-70. doi: 10.1001/jama.285.22.2864. PMID 11401607
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Background] Indredavik B, Rohweder G, Lydersen S. Frequency and effect of optimal anticoagulation before onset of ischaemic stroke in patients with known atrial fibrillation. J Intern Med. 2005 Aug;258(2):133-44. doi: 10.1111/j.1365-2796.2005.01512.x. PMID 16018790
- [Background] Saxena R, Lewis S, Berge E, Sandercock PA, Koudstaal PJ. Risk of early death and recurrent stroke and effect of heparin in 3169 patients with acute ischemic stroke and atrial fibrillation in the International Stroke Trial. Stroke. 2001 Oct;32(10):2333-7. doi: 10.1161/hs1001.097093. PMID 11588322
- [Background] Marini C, De Santis F, Sacco S, Russo T, Olivieri L, Totaro R, Carolei A. Contribution of atrial fibrillation to incidence and outcome of ischemic stroke: results from a population-based study. Stroke. 2005 Jun;36(6):1115-9. doi: 10.1161/01.STR.0000166053.83476.4a. Epub 2005 May 5. PMID 15879330
- [Background] Marfella R, Sasso FC, Siniscalchi M, Cirillo M, Paolisso P, Sardu C, Barbieri M, Rizzo MR, Mauro C, Paolisso G. Brief episodes of silent atrial fibrillation predict clinical vascular brain disease in type 2 diabetic patients. J Am Coll Cardiol. 2013 Aug 6;62(6):525-30. doi: 10.1016/j.jacc.2013.02.091. Epub 2013 May 15. PMID 23684685
- [Background] Hendrikx T, Hornsten R, Rosenqvist M, Sandstrom H. Screening for atrial fibrillation with baseline and intermittent ECG recording in an out-of-hospital population. BMC Cardiovasc Disord. 2013 Jun 10;13:41. doi: 10.1186/1471-2261-13-41. PMID 23758799
- [Background] Hendrikx T, Rosenqvist M, Sandstrom H, Persson M, Hornsten R. [Identification of paroxysmal, transient arrhythmias: Intermittent registration more efficient than the 24-hour Holter monitoring]. Lakartidningen. 2015 Jan 6;112:C6SE. Swedish. PMID 25584602
- [Background] Rizzo MR, Sasso FC, Marfella R, Siniscalchi M, Paolisso P, Carbonara O, Capoluongo MC, Lascar N, Pace C, Sardu C, Passavanti B, Barbieri M, Mauro C, Paolisso G. Autonomic dysfunction is associated with brief episodes of atrial fibrillation in type 2 diabetes. J Diabetes Complications. 2015 Jan-Feb;29(1):88-92. doi: 10.1016/j.jdiacomp.2014.09.002. Epub 2014 Sep 16. PMID 25266244
- [Background] Stamboul K, Zeller M, Fauchier L, Gudjoncik A, Buffet P, Garnier F, Guenancia C, Lorgis L, Beer JC, Touzery C, Cottin Y. Incidence and prognostic significance of silent atrial fibrillation in acute myocardial infarction. Int J Cardiol. 2014 Jul 1;174(3):611-7. doi: 10.1016/j.ijcard.2014.04.158. Epub 2014 Apr 22. PMID 24801093